CLINICAL TRIAL: NCT05229744
Title: Prevalence of Endolymphatic Hydrops in Patients With a History of Congenital Cytomegalovirus Infection With Symptomatic Cochleo-vestibular Involvement
Brief Title: Prevalence of Endolymphatic Hydrops With a Hitory of Congenital Cytomegalovirus Infection
Acronym: HYDROPS-CMV
Status: Terminated | Type: Observational
Why Stopped: The study was discontinued due to lack of inclusion.
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GPN_2021_23
Record Dates: First submitted 2021-09-29; First posted 2022-02-08 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Endolymphatic Hydrops
Keywords: CMV
MeSH Terms: conditions — Endolymphatic Hydrops

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: sequence MRI 3D FLAIR — Participation in this research entails the addition of an MRI sequence and an injection of contrast product (Gadovist®):
  - 3D FLAIR MRI sequence dedicated to the exploration of the inner ear, lasting 6min30s, performed 4 hours after the initial injection of contrast product

SUMMARY:
The management of patients with a history of congenital CMV infection (whether symptomatic or asymptomatic at birth) is modeled on their usual management.

DETAILED DESCRIPTION:
The management of patients with a history of congenital CMV infection (whether symptomatic or asymptomatic at birth) is modeled on their usual management.

Patients benefit as part of the care:

* A clinical cochleo-vestibular examination
* Functional otoneurological explorations: audiogram, caloric tests, vHIT, otolithic evoked potentials
* From an uninjected brain MRI

Participation in this research entails the addition of an MRI sequence and an injection of contrast product (Gadovist®):

- 3D FLAIR MRI sequence dedicated to the exploration of the inner ear, lasting 6min30s, performed 4 hours after the initial injection of contrast product.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 6 months old
* With a history of confirmed congenital CMV infection
* Suffering from symptomatic cochleo-vestibular dysfunction (average hearing threshold> 20dB in at least one ear and / or abnormal functioning of one or more sectors at the vestibular level)
* For adult patients, having received informed information about the study and having signed a consent to participate in the study
* For minor patients written consent of the two holders of the exercise of parental authority
* Affiliate or beneficiary of a social security scheme

Exclusion Criteria:

* Patient benefiting from a legal protection measure
* Pregnant or breastfeeding woman
* Contraindication to MRI (implanted electrical device, metallic foreign body, claustrophobia)
* Patient with a proven allergy to gadolinium
* Injection of gadolinium in the previous 7 days
* Known impairment of renal function ((estimated GFR <60 mL / min / 1.73 m²)

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a confirmed history of congenital CMV infection with symptomatic cochleo-vestibular dysfunction (mean hearing threshold> 20dB in at least one ear and / or functional abnormality in one or more areas at the vestibular level)
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2025-04-22 (Actual); Study Completion 2025-04-22 (Actual)

PRIMARY OUTCOMES:
the prevalence of at least one endolymphatic hydrops in patients with a history of congenital CMV infection with symptomatic cochleovestibular dysfunction | 4 hours after the initial injection of gadolinium, at least for one of the two ears
  Endolymphatic hydrops visualized with 3D FLAIR sequence in MRI

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hôpital Fondation Adolphe de Rothschild, Paris, PARIS
  - Hôpital Robert Debre, Paris

IPD SHARING:
Plan to Share IPD: No